CLINICAL TRIAL: NCT04024722
Title: Improving the Results of in Vitro Fertilization in Women With Poor Ovarian Response and Early Ovarian Insufficiency
Brief Title: Improving in Vitro Fertilization in Women With Poor Ovarian Response
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Barzilai Medical Center (Other)
Responsible Party: Principal Investigator, Shevach Friedler, Prof, Director of IVF unit, Barzilai Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0019-18-BRZ
Record Dates: First submitted 2019-07-03; First posted 2019-07-18 (Actual); Last update posted 2021-07-28 (Actual); Status verified 2021-07

CONDITIONS: Poor Ovarian Response; Ovarian Insufficiency
MeSH Terms: interventions — Fertilization in Vitro

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Single ovary treatment (Experimental)
  Interventions: Procedure: In Vitro Fertilization
- Dual ovary treatment (Experimental)
  Interventions: Procedure: In Vitro Fertilization

INTERVENTIONS:
Procedure: In Vitro Fertilization — Patients suitable for research with poor ovarian response will receive treatment including laparoscopic surgery, resection, and transplantation of ovarian tissue in the same operation to improve the chances of success of in vitro fertilization and pregnancy. Participants will be assessed for surgical incisions and fertility assessment up to two weeks after treatment, including general physical examination, US pelvic examination, and blood tests for a hormonal profile to determine the initiation of ovarian stimulation and IVF. Patients will be monitored from 2 weeks to 1 year after treatment (once a week in the first two months and one month for one year after surgery), which will include a general physical examination, a US test, and blood tests for the hormonal profile at the IVF clinic.

SUMMARY:
Improving the results of in vitro fertilization in women with poor ovarian response and early ovarian insufficiency

DETAILED DESCRIPTION:
BACKGROUND: Mechanical disruption of the Hippo signaling pathway in the ovaries can increase the likelihood of pregnancy and childbirth in women with early ovarian insufficiency. The method may also "work" in women with poor ovarian reserve and poor response to routine fertility treatments.

OBJECTIVE: To examine whether mechanical stimulation of ovaries by cutting the ovarian cortex treatment can increase eggs number aspirated during In Vitro Fertilization (IVF).

METHODS: Patients eligible for the study with poor ovarian response will receive treatment including laparoscopic surgery, resection, and transplantation of ovarian tissue in the same operation to improve the chances of IVF success and pregnancy. Participants will be assessed for surgical incisions and fertility assessment up to two weeks after treatment, including general physical examination, US pelvic examination, and blood tests for a hormonal profile to determine the initiation of ovarian stimulation and IVF. Patients will be monitored from 2 weeks to 1 year after treatment (once a week in the first two months and one month for one year after surgery), which will include a general physical examination, a pelvic ultrasound (US) and blood tests for the hormonal profile at the IVF clinic.

ELIGIBILITY:
Inclusion Criteria:

* Volunteers with poor ovarian response to standard fertility treatments according to the criteria of the European Fertility Association (ESHRE).
* Diagnosis of early ovarian insufficiency or symptoms that predict early ovarian insufficiency (imminent) seeking to become pregnant.

Exclusion Criteria:

Volunteers with

* Severe endometriosis diagnosed with laparoscopy.
* Previous major surgery involving ovaries.
* Ovarian cancer.
* Female reproductive malformations.
* Contraindications for laparoscopic surgery.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 40 (Estimated)
Dates: Start 2020-01-14 (Actual); Primary Completion 2021-07-31 (Estimated); Study Completion 2022-07-31 (Estimated)

PRIMARY OUTCOMES:
Number of oocytes | up to 1 year
  Number of oocytes
Fertilization rate | up to 1 year
  Fertilization rate
Embryos number | up to 1 year
  Embryos number
Pregnancies rate | up to 1 year
  Pregnancies rate

CONTACTS AND LOCATIONS:
Locations (1):
- Barzilay University Medical Center, Ashkelon, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Grin L, Berkovitz-Shperling R, Goldstein G, Michailov Y, Gemer O, Anteby E, Kawamura K, Saar-Ryss B, Friedler S. Drug-free in vitro activation of ovarian follicles and fresh tissue autotransplantation in patients with poor ovarian response and premature ovarian insufficiency. F S Sci. 2025 Aug;6(3):303-311. doi: 10.1016/j.xfss.2025.04.002. Epub 2025 Apr 30. PMID 40315958